CLINICAL TRIAL: NCT05660070
Title: Context-Aware Mobile Intervention for Social Recovery in Serious Mental Illness
Acronym: mSITE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Eric Granholm, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R61MH126094 (NIH)
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Mood Disorder, Psychotic
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Affective Disorders, Psychotic

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mobile Social Interaction Therapy by Exposure (mSITE) (Experimental): mSITE is a blended intervention that integrates brief in-person psychotherapy with context-triggered mobile smartphone intervention and remote telephone coaching.
  Interventions: Behavioral: mobile Social Interaction Therapy by Exposure (mSITE)

INTERVENTIONS:
Behavioral: mobile Social Interaction Therapy by Exposure (mSITE) — mSITE is a blended intervention that integrates brief in-person psychotherapy with context-triggered mobile smartphone intervention and remote telephone coaching.

SUMMARY:
This open trial will test a new technology-supported blended intervention, mobile Social Interaction Therapy by Exposure (mSITE), that targets social engagement in consumers with serious mental illness.

DETAILED DESCRIPTION:
Social isolation is common in serious mental illness and has a profound negative impact on recovery. This study evaluates a new technology-supported blended intervention, mobile Social Interaction Therapy by Exposure (mSITE), that targets social behavior, and it also validates several new techniques for measuring social behavior. mSITE blends brief in-person psychotherapy with context-triggered mobile smartphone intervention and remote telephone coaching. The investigators will conduct an open trial of mSITE, evaluating whether the intervention leads to clinically significant changes in the frequency of social interactions. The investigators will also determine the dose of app plus remote coaching necessary to achieve this effect, by evaluating change at 12, 18, or 24 weeks. If found to be effective, a scalable intervention that reduces social isolation in serious mental illness would have significant personal, societal, and economic impact.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary informed consent to participate and capacity to consent;
2. Age 18 to 65;
3. DSM-5 diagnosis of schizophrenia, schizoaffective, bipolar I disorder or major depression with history of psychosis based on a SCID-5 interview and available medical record review;
4. Minimum level of social avoidance defined by a score of ≥ 2 on the Scale for the Assessment of Negative Symptoms (SANS) asociality item;
5. ≥ 6th grade reading level on the Wide Range Achievement Test-4 Reading subtest (to read therapy workbook).

Exclusion Criteria:

1. Prior CBT in the past 2 years;
2. Greater than moderate disorganization on the PANSS (P2- Disorganization item >5);
3. DSM-5 alcohol or substance dependence in past 3 months based on the SCID;
4. Level of care required interferes with outpatient therapy (e.g., hospitalized; severe medical illness)
5. Unable to adequately see or manually manipulate a phone;
6. Resident of an integrated housing facility that also provides treatment services.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

PRIMARY OUTCOMES:
Ecological Momentary Assessment | Assess change from baseline in number of social interactions at Weeks 0, 8, 12, 18, and 24
  EMA is a method of remote data collection that involves repeatedly sampling a participant's current behaviors, thoughts, mood, and experiences in real time, in their natural environments. The primary outcome in this study will be the number of social interactions.
Clinical Assessment Interview for Negative Symptoms | Assess change from baseline in expression and motivation and pleasure at Weeks 0, 8, 12, 18, and 24
  Measure changes in motivational negative symptoms on the CAINS. The CAINS is a 13-item interview-based assessment of negative symptoms, and each item is rated from 0 (no impairment) to 4 (severe deficit) measuring the two negative symptom factors recommended in consensus reports: Expression and Motivation and Pleasure (MAP) across social, vocational and recreational domains. Total scores for each factor are computed. The range for the MAP is 0 - 36, and the range for the Expression factor is 0 - 16. Higher scores indicate more severe negative symptoms for both factors.
Birchwood Social Functioning Scale | Assess change from baseline in social functioning at Weeks 0, 8, 12, 18, and 24
  Measure changes in functioning on the Birchwood Social Functioning Scale (SFS). The SFS is a self-report assessment of functioning with 7 subscales, and each item is rated from 0 to 3 with the exception of the Occupation/Employment subscale if a participant is in regular employment (scores range from 7-10 based upon type of work). The subscales and score ranges are: Social Engagement Withdrawal (0-15), Interpersonal Communication/Relationships (0-30), Prosocial Activities (0-66), Recreation (0-48), Independence-Performance (0-39), Independence-Competence (0-39), and Occupation/Employment (0-10). Higher scores indicate better functioning for all subscales.
Positive And Negative Syndrome Scale | Assess change from baseline in positive and negative symptoms at Weeks 0, 8, 12, 18, and 24
  The PANSS is a 30-item interview that provides balanced representation of positive and negative symptoms and gauges their relationship to one another and to global psychopathology. Items are rated 1 (Absent) to 7 (Extreme) and summed across items for a total range of scores of 30-210. Higher scores indicate the presence of more severe symptoms.
Passive sensing mobile application | Assess change from baseline in number of conversations at Weeks 0, 8, 12, 18, and 24
  The passive sensing mobile application will measure the number of conversations. The conversations or specific content will not be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Granholm, PhD, Principal Investigator — University of California, San Diego; San Diego Veterans Healthcare System
Locations (1):
- UC San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Per terms of the award, participant-level data will be uploaded to the NIMH Data Archive (NDA).
Time Frame: Data will be uploaded according to NDA standard data submission periods. These periods are currently twice each year.
Access Criteria: Data access is outlined in the current NDA Policy.
URL: https://nda.nih.gov/

DOCUMENTS (1):
  • Informed Consent Form (2023-01-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT05660070/ICF_001.pdf